CLINICAL TRIAL: NCT05197491
Title: Recognizing Menstrual Disturbance During COVID-19 Pandemic Among Obstetrics and Gynecology Healthcare Professionals, Fayoum University Hospital.
Brief Title: Women's Menstruation During the Covid-19 Pandemic
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, rehab abdelhamid aboshama, lecturer of obstetrics and gynecology Faculty of medicine, Fayoum University
Other Study IDs: R 179
Record Dates: First submitted 2022-01-07; First posted 2022-01-19 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Menstrual Irregularity; Stress Related Disorder; COVID-19 Pneumonia; Fear; Anxiety
Keywords: COVID-19; Work-related stress; Health care worker; Survey; Menstrual irregularity
MeSH Terms: conditions — Menstruation Disturbances; Anxiety Disorders; COVID-19; Occupational Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The COVID-19 crisis has rapidly become the most significant public health crisis of our times. It has particularly impacted healthcare workers (HCW) due to the over-whelming of healthcare resources, as well as a critical absence of protective equipment and risk to their own health as well as the risk of exposure to their family. All these factors have likely resulted in significant levels of stress, anxiety, and affection of the general health

DETAILED DESCRIPTION:
During the first wave of the pandemic, overstretched healthcare systems left health workers in hard-hit countries struggling with long working hours, fatigue, and extreme psychological stress. Rapidly vanishing supplies, national lockdown, and a feeding frenzy on the open market for personal protective equipment (PPE) led to shortages. Healthcare workers often had to care for patients with suspected or confirmed COVID-19 infection without proper training or adequate PPE. This contributed to an increased risk to healthcare workers during the initial phase of the pandemic.

Study Methods:

This is a retrospective cross-sectional study that will be conducted among healthcare professionals working in the obstetrics and gynecology department, Fayoum University Fayoum, Egypt. A survey-based study will be conducted between January 15 and March 1, 2022, using the database of Fayoum University. A self-administered online survey consisting of 80 questions was developed.

ELIGIBILITY:
Inclusion Criteria:

* All obstetrics and gynecology department healthcare workers who were or had been resident, physicians or consultant physicians, nurses, and paramedical healthcare active during the COVID-19 pandemic period at a designated Fayoum university hospital, regardless of gender, age, experience, and duration of employment.

Exclusion Criteria:

* Exclusion criteria:

  1. physicians who were retired or did not currently work in a designated COVID-19 hospital.
  2. Physicians from other specialties
  3. Physicians were on leave during the pandemic for various reasons.

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: A COVID-19 survey in electronic or hard copy format for healthcare workers include physicians, nurses, emergency medical personnel, medical and nursing students, and administrative staff.
  The survey included questions about the respondents' demographic characteristics, changes in their practice during the pandemic period, and basic knowledge of COVID-19. Furthermore, questions evaluating fear and stress associated with the pandemic. In addition, the change in the character of the menstrual cycle and sexual life.
  The participants will be informed that the survey will be intended for research and that their participation will be anonymous. Participants did not have to answer all the questions in order to complete the survey.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Rate of irregular menstrual cycle | 6 month after working in the pandemic
  Irregular menstrual cycle
Length of cycle | 6 month after working in the pandemic
  Length of cycle (days)
Rate of prolonged bleeding per cycle | 6 month after working in the pandemic
  Duration of bleeding (day)
Amount of flow | 6 month after working in the pandemic
  Number of used tampons (pads) during bleeding
Rate of dysmenorrhea | 6 month after working in the pandemic
  Dysmenorrhea status
Recognizing the stress related to work in the Covid-19 pandemic | 6 month after working in the pandemic
  The person is asked to answer the questions on the scale over the symptoms she has experienced during the past year including today'. Each item scores between 0 and 3 as none, mild, moderate, and severe, respectively.
Recognizing a change in sexual life | 6 month after working in the pandemic
  The participants will answer the survey by yes or no.

SECONDARY OUTCOMES:
The number of differences in menstrual cycle length | 6 month after working in the pandemic
  Menstrual cycle difference between Covid-19 positive and negative healthcare workers (days)
The number of differences in bleeding days | 6 month after working in the pandemic
  Duration of bleeding difference between covid positive and negative healthcare workers (days)
The number of differences in the amount of flow | 6 month after working in the pandemic
  Amount of flow difference between covid positive and negative healthcare workers (tampons)

CONTACTS AND LOCATIONS:
Locations (1):
- Fayoum university, Al Fayyum, Egypt

IPD SHARING:
Plan to Share IPD: No